CLINICAL TRIAL: NCT01982643
Title: CTN-0054 Accelerated Development of Additive Pharmacotherapy Treatment (ADAPT) for Methamphetamine Use Disorder
Brief Title: Accelerated Development of Additive Pharmacotherapy Treatment for Methamphetamine Use Disorder
Acronym: ADAPT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Walter Ling (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Walter Ling, Professor of Psychiatry and Director, UCLA Integrated Substance Abuse Programs, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0054; U10DA013045 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-13 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Methamphetamine Use Disorder
MeSH Terms: interventions — Naltrexone; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- naltrexone plus bupropion (Experimental): extended-release depot naltrexone (XR-NTX; as Vivitrol®)plus extended-release bupropion tablets (BRP; as Wellbutrin XL®)
  Interventions: Drug: naltrexone plus bupropion

INTERVENTIONS:
Drug: naltrexone plus bupropion — Participants will receive a monthly injection of extended-release depot naltrexone (XR-NTX; as Vivitrol®) plus once-daily bupropion extended-release tablets (BRP; as Wellbutrin XL®) for 8 weeks.

SUMMARY:
The aim of this 2-stage, 3-site study is to investigate the effectiveness and safety of a combination of extended-release depot naltrexone plus extended-release bupropion as a potential pharmacotherapy for methamphetamine (MA) use disorder.

DETAILED DESCRIPTION:
Stage 1 will include 20 individuals with severe stimulant use disorder (methamphetamine type) enrolled across three study sites. Following a maximum 30-day screening period to establish eligibility, participants will receive a monthly injection of extended-release depot naltrexone (XR-NTX; as Vivitrol®) plus once-daily bupropion extended-release tablets (BRP; as Wellbutrin XL®) for 8 weeks. Take-home oral study medication (BRP) will be dispensed weekly for dosing on non-clinic days. Participants will be asked to attend clinic twice weekly for observed BRP dosing, collection of urine samples, assessments, and medical management. Following the 8-week active medication phase, participants will complete a follow-up phase, including a medication taper and post-medication phase follow-up visit during Week 9. If Stage 1 data document success (see criteria below) in at least 3 "responder" study participants, Stage 2 will follow utilizing the same protocol as in Stage 1, to enroll an additional group of 29 participants. Using the same criteria of "responder" success, if the combined stages document success in at least 9 of 49 study participants, the combination medication will be considered to have shown sufficient potential to advance to a large-scale placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 65 years of age;
* Be able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study;
* Demonstrate understanding of study procedures by correctly answering all questions on the consent competency tool;
* Be interested in reducing or stopping methamphetamine use;
* Meet DSM-5 criteria for severe methamphetamine use disorder;
* Meet subjective and objective methamphetamine use criteria as defined by the protocol;
* Meet subjective and objective measures of being opioid-free prior to enrollment and medication induction per study medical clinician's determination (including passing a naloxone challenge);
* Agree to use study cellphone to record videos of take-home dosing for transfer to study team.
* If female of childbearing potential, agree to use acceptable birth control methods during participation in the study;

Exclusion Criteria:

* Have known allergy or sensitivity to study medications;
* Have a medical history or condition that would make study participation difficult or unsafe;
* Have an acute psychiatric disorder or condition that would make study participation difficult or unsafe;
* Liver function test results greater than 5 times the upper limit of normal or other exclusionary clinical lab test values;
* Recent or ongoing treatment with medications that, in the judgment of the study medical clinician, could interact adversely with study drugs or interfere with study participation;
* Have a current pattern of alcohol, benzodiazepine, or other sedative-hypnotic use, as determined by the study medical clinician, which would preclude safe participation;
* Pending action or situation that might prevent remaining in the area for the duration of the study or prevent participation in study activities
* Be currently pregnant or breastfeeding;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — UCLA Integrated Substance Abuse Programs; Larissa Mooney, M.D., Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (3):
- United States (3):
  - UCLA Integrated Substance Abuse Programs, Los Angeles, California
  - University of Hawaii, Honolulu, Hawaii
  - Nexus Recovery Center, Dallas, Texas

REFERENCES:
- [Derived] Walker R, Hillhouse M, Perrochet B, Sparenborg S, Mooney L, Ling W. Medication Adherence Monitoring Using Smartphone Video Dosing in an Open-label Pilot Study of Monthly Naltrexone Plus Once-daily Bupropion for Methamphetamine Use Disorder: Feasibility and Acceptability. J Addict Med. 2019 Sep/Oct;13(5):372-378. doi: 10.1097/ADM.0000000000000509. PMID 30724759
- See also: NIDA Clinical Trials Network Dissemination Library — http://ctndisseminationlibrary.org/
- See also: NIH National Institute on Drug Abuse Clinical Trials Network — http://www.drugabuse.gov/CTN
- See also: UCLA Integrated Substance Abuse Programs (ISAP) — http://www.uclaisap.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone Plus Bupropion
Started | 49
Completed | 37
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Naltrexone Plus Bupropion
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Participants Categorized as "Responders"
Description: Study "Responders" were defined as participants providing six MA-negative urine tests of eight administered in the evaluation period (the last four weeks of the active medication phase), including the last test collected in the final study week of the active medication phase.
Time Frame: Weeks 4-8
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone Plus Bupropion
Number analyzed (Participants) | 49
Participants | 11

ADVERSE EVENTS:
Arm/Group | Naltrexone Plus Bupropion
Serious Adverse Events (participants affected / at risk) | 2/49
Other Adverse Events (participants affected / at risk) | 45/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone Plus Bupropion (N=49)
Inpatient admission to hospital or prolongation of existing hospitalization (Surgical and medical procedures) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone Plus Bupropion (N=49)
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 3
Nasopharyngitis (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 5
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Fatigue (General disorders) | 4
Irritability (General disorders) | 3
Hyperthyrodism (Vascular disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Couth (Respiratory, thoracic and mediastinal disorders) | 3
Tachycardia (Cardiac disorders) | 6
Vision blurred (Eye disorders) | 4
Decreased appetitite (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No